CLINICAL TRIAL: NCT02463539
Title: Residual Anti-pneumococcal Immunity After Pneumococcal Immunization in ANCA-associated Vasculitis. PneumoVas Pilot 1
Brief Title: Residual Anti-pneumococcal Immunity After Pneumococcal Immunization in ANCA-associated Vasculitis
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI 15001
Record Dates: First submitted 2015-05-12; First posted 2015-06-04 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Pneumococcal Infection; ANCA-associated Vasculitis
Keywords: Pneumococcal infection; Invasive pneumococcal disease (IPD); Pneumococcal vaccine; Systemic vasculitis; ANCA-associated vasculitis; Vaccinology; Immunocompromised; Auto-immune disease
MeSH Terms: conditions — Pneumococcal Infections; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Systemic Vasculitis

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

SUMMARY:
Descriptive study of the residual anti-pneumococcal immunity in patients with Anti-neutrophil cytoplasmic antibody (ANCA)-associated vasculitis (AAV) who have previously gone through pneumococcal immunization.

DETAILED DESCRIPTION:
The purpose of this study is to determine, through serotype-specific enzyme linked immunosorbent assay (ELISA) and opsonophagocytosis (OPA) titres whether AAV patients who have gone through pneumococcal vaccination are protected against invasive pneumococcal diseases (IPD).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Anti-neutrophil cytoplasmic antibody (ANCA)-associated vasculitis: diagnosis for granulomatosis with polyangiitis, microscopic polyangiitis or eosinophilic granulomatosis with polyangiitis according to American College of Rheumatology criteria
* Anti-pneumococcal immunization in the past 36 months
* History of anti-pneumococcal vaccination according to French recommendations (simple vaccine schedule with PPV23 or combine vaccine schedule with PCV13 followed by PPV23 8 weeks later)

Exclusion Criteria:

* Known or suspected pregnancy
* Splenectomy
* Patient without social security coverage
* Patient opposal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed for Anti-neutrophil cytoplasmic antibody (ANCA)-associated Vasculitis
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2015-09; Primary Completion 2015-12 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Residual anti-pneumococcal immunity after pneumococcal immunization. | visit V0 (day 0)
  Proportion of patients at baseline (V0) with ≥1 µg/mL ELISA immunoglobulins G (IgG) antibody titers to at least 6 of the 10 shared serotypes (i.e. 3, 4, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F) included both in the 13-valent conjugate pneumococcal vaccine (PCV13) and in the 23-valent non-conjugate pneumococcal vaccine (PPV23)

SECONDARY OUTCOMES:
To assess serotype 3, 4, 6B, 7F, 9V, 14, 18C, 19 A, 19F, 23F, 10A and 12F-specific residual immunity after vaccination | visit V0 (day 0), visit V-1 (pre immunization)
  ELISA specific antibody titres to serotype 3, 4, 6B, 7F, 9V, 14, 18C, 19 A, 19F, 23F (included both in PCV13 and PPV23), 10A and 12F (specific to PPV23)
For each of the following serotypes (3, 4, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F), to assess among ELISA-protected patients (i.e. with a ≥1 µg/mL ELISA IgG antibody titer) the proportion who also show in vitro opsonophagocytic antibody activity | visit V0 (day 0)
  Descriptive analysis:
  a/ For each of the following serotypes (3, 4, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F), opsonophagocytosis (OPA) titers will be measured in ELISA-protected patients at V0. Opsonophagocytic antibody activity is considered positive if the antibody titer is above a serotype-specific predefined threshold.
  B/ The proportion of overall OPA-protected patients (meaning ≥ 50% of OPA positive serotypes )
For patients for whom pre-vaccinal serum is available (via the PHENOVASC bank), to assess the impact of immunization on serotype-specific ELISA antibody titer and OPA activity. | visit V-1 (pre immunization) ; visit V0 (day 0)
  For patients already included in the PHENOVASC study (V-1) ≤6 months before receiving pneumococcal immunization, anti-pneumococcal immunity will be assessed for serotype 3 , 4 , 6B, 7F, 9V, 14 , 18C, 19A , 19F , 23F, 10A and 12F (with ELISA only for the two latter).
  For each serotype:
  In ELISA, we will describe the proportion of responding patients (i.e. with a two-fold increase from V-1 to VO and a ≥1 μg/ml titre at V0.
  In VO ELISA-responding patients, OPA titers will be measured. An opsonophagocytic antibody activity is considered positive if the antibody titer shows a four-fold increase from V-1 to V0 and is above a serotype-specific predefined threshold.
Composite Outcome Measures - To identify epidemiologic, clinic and biologic predictive factors that may influence vaccine-induced immune response. | visit V-1 (pre immunization) ; visit V0 (day 0)
  Analysis of epidemiological, clinical and biological data collected during follow-up: age, sex, history of immunosuppressive therapy, time since previous PPV23 injection, number of previous PPV23 immunizations, AAV activity and severity according to Birmingham Vasculitis Activity Score and Vasculitis Damage Index, results of biological analyses

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu Groh, MD, MSc, Principal Investigator — AP-HP- Cochin hospital
Locations (1):
- AP-HP ; Cochin Hospital, Paris, Île-de-France Region, France